CLINICAL TRIAL: NCT07009886
Title: Development of an Educational Patient Decision Aid (Treatments in Advanced Cancer - Decision Aid, TA-DA) to Promote Shared Decision Making for Third-line or Beyond Palliative Systemic Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-0480; NCI-2025-03797 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TA-DA (Experimental): Patient and caregiver participants are presented with a prototype version of TA-DA and participate in interviews over 90 minutes to further refine the tool.
  Interventions: Other: Communication
- EUC (Experimental): Patient and caregiver participants are presented with a prototype version of TA-DA and participate in interviews over 90 minutes to further refine the tool.
  Interventions: Other: Communication

INTERVENTIONS:
Other: Communication — Participants meet with clinician

SUMMARY:
To develop an educational patient decision aid for advanced cancer patients to prepare them to have conversations with their clinicians about treatment options (Treatments in Advanced cancer - Decision Aid, TA-DA).

DETAILED DESCRIPTION:
Primary Objectives:

The study objective is to develop an educational patient DA (Treatments in Advanced cancer - Decision Aid, TA-DA) to assist patients, their caregivers, and clinicians to make an informed decision about third-line or beyond palliative systemic therapy for advanced cancer. To fulfill the study's objectives, we will complete 3 study parts:

Using qualitative methods, explore the decision-making needs of patients with advanced cancer, their caregivers, and clinicians, about third-line or beyond palliative systemic therapy; identify initial preferences and recommendations to inform the design of the educational patient DA in Part II.

Following a user-centered design approach, develop and measure the acceptability of an educational patient DA to promote shared decision making among patients with advanced cancer, their caregivers, and clinicians, about third-line or beyond palliative systemic therapy.

Conduct a pilot RCT to estimate the effect of the educational patient DA (TA-DA) on patient's knowledge of their treatment options.

Secondary Objectives:

Examine the impact of the educational patient DA (TA-DA) on patients' illness understanding (Prigerson's items), preparation for decision making (PrepDM Scale), decisional conflict (Decisional Conflict Scale [DCS]), quality of the shared decision-making process (SDM Process Scale), decisional regret (decisional regret scale), therapeutic alliance (The Human Connection Scale [THC]), anxiety (Generalized Anxiety Disorder 7 [GAD-7]), final treatment choice, and end-of-life care outcomes (e.g., systemic therapy use in last month of life).

Examine the impact of the educational patient DA (TA-DA) on caregivers' knowledge of the patient's treatment options, illness understanding (Prigerson's items), preparation for decision making (PrepDM Scale), decisional conflict (DCS), quality of the shared decision- making process (SDM Process Scale), therapeutic alliance (THC Scale), and anxiety (GAD-7).

Examine the acceptability (Ottawa Acceptability Scale) of the educational patient DA (TA-DA) among patients, caregivers, and oncologists in the educational patient DA group. Examine the acceptability (modified Acceptability of Intervention Measure [AIM]), appropriateness (Intervention Appropriateness Measure [IAM]), and feasibility (Feasibility of Intervention Measure [FIM]) of the educational patient DA (TA-DA) among clinicians in the educational patient DA group.

Exploratory Objective:

2.3.1. (Part III) Examine the impact of the educational patient DA (TA-DA) on the concordance between patient-caregiver dyads for knowledge of the patient's treatment options, illness understanding (Prigerson's items), preparation for decision making (PrepDM Scale), decisional conflict (DCS), quality of the shared decision-making process (SDM Process Scale), therapeutic alliance (THC Scale), and anxiety (GAD-7).

ELIGIBILITY:
Inclusion Criteria:

1. Clinicians (Part I/II/III):

   MD Anderson medical oncologists and APPs who provide care to patients with advanced cancer
2. Patients (Part I/II/III):

   Age 18 or over
   * Diagnosis of advanced cancer (i.e., metastatic, relapsed, and/or incurable disease as defined by the treating oncologist) who has received at least 2 lines of palliative systemic therapy*
   * Patient-rated ECOG performance status of 1-3 for Part I/II and 2-3 for Part III
   * Able to make treatment decisions based on the clinical judgement of the oncology team
   * English speaking

     * patient has started, is receiving, and/or has completed second-line palliative systemic therapy or beyond
3. Caregivers (Part I/II/III):

   * Age 18 or older
   * Currently a primary caregiver to a patient who satisfies the patient eligibility criteria listed above
   * For the study purposes, a primary caregiver is defined as:

     * someone who provides physical, emotional, decisional and/or logistical assistance to the patient regularly (e.g. daily, weekly);
     * can be a family member, friend, or other individual in a close relationship with the patient;
     * must be identified by the patient and self-identify as the primary person providing caregiving support to the patient
   * Able to provide informed consent and participate in the study
   * English speaking

Exclusion Criteria:

Any patient who meets any of the following criteria will be excluded from participation in this study:

* (Part I/II/III): Diagnosis of cognitive impairment or dementia requiring a surrogate decision maker as determined by the clinical team
* (Part III only): Participants in Part I and II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org